CLINICAL TRIAL: NCT02432222
Title: Effects of Visual Arts Training on Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: York University (Other)
Responsible Party: Principal Investigator, Melody Wiseheart, Associate Professor, York University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YorkU-AD1
Record Dates: First submitted 2015-04-01; First posted 2015-05-04 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Dementia; Alzheimer Disease
MeSH Terms: conditions — Dementia; Alzheimer Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Music Training (Experimental): Music training
  Interventions: Behavioral: Music Training
- Visual Arts Training (Experimental): Visual arts training
  Interventions: Behavioral: Visual Arts Training
- Control (No Intervention): Waitlist control

INTERVENTIONS:
Behavioral: Visual Arts Training — Visual arts training
  Arms: Visual Arts Training
Behavioral: Music Training — Music training
  Arms: Music Training

SUMMARY:
The study will use a randomized controlled trial to test the efficacy of two interventions (visual arts and music) for individuals with dementia, focusing on dementia of the Alzheimer's type (DAT). Interventions will be run for 10 weeks in dementia day centers and/or retirement residences. Participants will be tested before and after the intervention on a battery of cognitive, affective, and behavioural measures. They will be compared to a waitlist control group who don't receive the intervention.

The purpose of our research is twofold: treatment of symptoms and improved quality of life during disease progression in dementia. For the primary aim, the investigators are examining the potential of arts interventions on declining functions in dementia (memory, mood, and behavior) to investigate potential treatment effects. Secondly, quality of life will be measured, with the aim of looking beyond disease progression to contribute to an overall positive patient experience. Research has indicated the need for non-pharmacological treatments to be used as a first line of action against dementia symptoms and development. While, in best practice, pharmacological treatments should be used as a second-line approach.

Note: Music intervention dropped prior to study initiation.

DETAILED DESCRIPTION:
Participants

Older adults age 65 and older, both males and females, with normal or corrected vision and hearing. Participants will require a diagnosis of dementia, with no other known comorbid cognitive or neurological impairments.

Participants will be randomly allocated to one of three groups

1. Visual arts intervention group
2. Music intervention group
3. Waitlist control group (receiving the intervention after the completion of both testing sessions).

Data analysis

1. Mixed 2x3 analysis of variance (ANOVA) for each construct, with within-subject factor of time (pre-intervention and post-intervention) and between-subject factor of group (visual arts, music, control).
2. Test for confounding effects of background factors (socioeconomic status, education level, gender, activity participation).
3. Mediation analyses for effects of mood on cognition and behaviour.

Procedure

The present study is a randomized controlled trial assessing three groups of dementia patients: a visual art group, a music group, and a non-art waitlist control group. Randomized control trials are needed in dementia research because few experimental studies exist to support that training has a causal influence on dementia related decline. Older adults with dementia will be allocated to either a visual art group, music group, or waitlist control group. Using two arts forms enables us to have active control groups to examine the specificity of observed effects.

To address inconsistencies and methodological issues in existing results, the current study will use rigorous experimental control, such as allocation concealment, adequate sample size, and tester blinding. Based on a power calculation using effect sizes from previous studies, each group will have sixty participants for an adequately powered sample. Participants will be recruited by contacting activity administrators at dementia retirement residences and day programs. Attention has and will be taken to prevent attrition, such as tailoring interventions towards participants' needs and capacities, and by involving families and caregivers in the research. Furthermore, the intervention and assessments will be conducted at the participant's respective care facility. Currently, the investigators have an established partnership with day dementia programs in the Toronto area, and will be negotiating agreements to work with other senior retirement residences and day programs. Recruiting from multiple locations and randomly assigning participants to experimental or control groups will help with generalizability of results.

Following previous studies, the art interventions will take place over ten weeks (one hour per day, two days per week). The visual art course will be a drawing course focusing on basic visual art concepts (such as shape and contrast) and the music course will be a singing and instrumental course focusing on basic music concepts (such as rhythm and melody). Defining training elements will delineate the specific effects of different activities on cognition, a poorly explored area in previous studies. The visual arts and music courses will be taught by the study's graduate student investigators (Annalise D'Souza and Katherine Matthews). Both teachers have experience and accreditations in their respective art.

Before and after both courses, all participants (wait-list control group included) will complete multiple assessment tasks. Data will be analyzed using mixed analyses of variance to compare performance for each participant at both testing sessions, and between groups. The pre-tests will occur one to two weeks before the beginning of the arts courses, and the post-tests will occur during the two weeks after the art courses are finished. Testing will occur over a two day period, for one hour per day to accommodate participants attention span and cognitive load. All tasks have been selected for their reliability, validity, and their suitability to the population at hand. To investigate specific influences of each art, separate visual and auditory/verbal tests will be used for each measure. Testing and courses will begin in early 2015, and will be run multiple times at different locations to reach the targeted sample size, with expected start dates in April, September, and January. Participant recruitment for these courses will begin in April and continue until December. Based on previous discussions with dementia day programs, and the attrition and admission rates of these programs, attaining sixty participants per group by December will be possible if the investigators continue recruiting from multiple day programs and retirement residences.

The participants' involvement in the study is completely voluntary and the participant and their caregiver (if substitute consent is required) may choose to stop their participation at any time. In the event the participant withdraws from the study all associated collected data will be immediately destroyed wherever possible. All information the participant supplies during the study will be held in confidence. Confidentiality will be provided to the fullest extent possible by law.

Hypotheses

Predictions are outlined in the hypotheses below:

1. Visual art and music training will offset some of the decline in cognitive functions (working memory, long-term memory, selective attention, dual-tasking, and task switching).

   a. Effects of visual art will be greater on visual measures of cognition and effects of music will be greater on auditory measures
2. Visual art and music training will improve mood and lessen problematic behavior.
3. Visual art and music training will improve overall quality of life.
4. Mood will mediate some of the changes in cognition and behaviour

Background

The present study focuses on non-pharmacological art interventions for persons with Alzheimer's disease and related dementias. Arts interventions will be designed and implemented to investigate the effects of arts training on disease symptomology and overall quality of life for persons with dementia. Dementia can be characterized by declining cognitive functions, accompanied by a loss of daily functioning (DSM-IV, 2000), with a range of cognitive, behavioural, and psychological deficits for different types of dementia.

The study will use a randomized controlled trial to test efficacy of two arts interventions. Arts and dementia experts will guide intervention design to ensure that programs are powerful and controlled. With the aims of reliability and applicability, interventions will be created that can be tested by future researchers and applied by real-world practitioners. Effects will be evaluated with a broad range of measures (affective, cognitive, and behavioural. The proposed study is significant for two reasons. First, it addresses a repeatedly highlighted need for non-pharmacological interventions in treating dementia. Second, it looks beyond disease treatment alone by looking to also improve overall quality of life in patients with dementia.

Non-pharmacological interventions offer great potential for mental improvement, but further experimental research is needed before efficacy is established. A large evidence base demonstrates a cognitive benefit of arts on healthy older adults. It is uncertain however, whether such findings also apply to individuals with dementia. A few preliminary studies indicate similar benefits can be found, but not all studies have reported cognitive improvements following arts interventions in this patient population. In addition, prospective studies indicate a link between dementia and cognitively stimulating activities such as the arts. For example, it has been supported that older adults who participate in more stimulating activities also display fewer incidences of dementia and Alzheimer's disease.

Research suggests that non-pharmacological treatments should be used as a first line of action against dementia, while pharmacological treatments should serve as a second-line approach. While non-pharmacological treatments have indicated remedial effects, there is a need for reliably conducted experiments to establish efficacy. Art recreation is easy to administer, inexpensive and non-time consuming. Unlike the majority of current pharmacological treatments, it is a noninvasive and pleasurable activity, and maintains the personhood of the individual with dementia.

Note: Music intervention dropped prior to study initiation, due to insufficient participant recruitment.

ELIGIBILITY:
Inclusion Criteria:

* dementia

Exclusion Criteria:

* known comorbid cognitive or neurological impairments

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 23 (Actual)
Dates: Start 2015-04; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment (MOCA, change measure) | baseline and 8 weeks
  Designed by Nasreddine (2005) for overall cognitive assessment
Working memory (change measure) | baseline and 8 weeks
  Visual (body part pointing test, Stopford et al, 2010), auditory (digit span test, Weschler, 2008)
Rey-Osterreith test of long-term memory (change measure) | baseline and 8 weeks
  Rey-Osterreith Complex Figure Recognition, Rey-Osterreith Figure Copy, Rey-Osterreith verbal task (Osterreith, 1944; Schmidt, 1996)
Trails test of set-shifting (change measure) | baseline and 8 weeks
  Measure of set-shifting/task switching
Dual task for visual and auditory search (change measure) | baseline and 8 weeks
  designed by Baddeley (2001)

SECONDARY OUTCOMES:
Behavioural psychiatric peformance (time-to-event measure) | from date of randomization upto 8 weeks
  Neuropsychiatric Inventory (NPI; Cummings, 2009)
Quality of Life (change measure) | baseline and 8 weeks
  Questionnaire on well-being (Kerner, Patterson, Grant, & Kaplan, 1998) to be filled out by caregivers
Visual analog mood scale | baseline and 8 weeks
  Measure of mood designed by Stern et al (2010) and Temple et al (2004)

CONTACTS AND LOCATIONS:
Overall Officials: Melody Wiseheart, PhD, Principal Investigator — York University

IPD SHARING:
Plan to Share IPD: Undecided